CLINICAL TRIAL: NCT00344006
Title: A Multi-centre, Randomised, Double-blind, Double Dummy Study Comparing the Efficacy and Safety of Chlorproguanil-dapsone-artesunate Versus Artemether-lumefantrine in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Children and Adolescents in Africa.
Brief Title: Chlorproguanil-Dapsone-Artesunate Versus COARTEM For Uncomplicated Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDA 714703/005
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Malaria, Falciparum
Keywords: Malaria CDA COARTEM Africa pediatrics children
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: chlorproguanil-dapsone-artesunate; Drug: artemether-lumefantrine

INTERVENTIONS:
Drug: chlorproguanil-dapsone-artesunate
Drug: artemether-lumefantrine
  Other Names: chlorproguanil-dapsone-artesunate

SUMMARY:
Chlorproguanil-dapsone has been approved for the treatment of uncomplicated Plasmodium falciparum malaria in a number of countries across sub-Sahara Africa, and by the UK's Medicines and Healthcare products Regulatory Agency.

CDA is a combination of chlorproguanil, dapsone and artesunate, being developed in a public-private partnership with the Medicines for Malaria Venture (MMV), World Health Organisation (WHO-TDR) and academic partners from the London School of Hygiene and Tropical Medicine, University of Liverpool and the Liverpool School of Tropical Medicine as a treatment for acute uncomplicated P. falciparum malaria.

The combination of chlorproguanil-dapsone-artesunate (CDA) is being developed to supersede chlorproguanil-dapsone for the same indication, but the addition of an artemisinin derivative, artesunate, should provide additional population benefits over chlorproguanil-dapsone alone. The artemisinins have been demonstrated to rapidly reduce parasite load and have activity against the sexual stages of the P.falciparum lifecycle. The addition of a second agent to the chlorproguanil-dapsone combination should also protect against the selection of resistant strains of P.falciparum.

Artemether-lumefantrine is the only available fixed-dose Artemisinin-based Combination Therapy actually available and is considered as the gold standard for the treatment of P. falciparum malaria. This study will therefore aim to demonstrate the non-inferiority of the combination of CDA to artemether-lumefantrine in terms of efficacy at 28-days. The key secondary objectives will compare the Parasite Clearance Times (PCT) and the Fever Clearance Times (FCT) between CDA and artemether-lumefantrine.

ELIGIBILITY:
Inclusion criteria:

* Acute, uncomplicated P.falciparum malaria, microscopically confirmed
* Temperature at screening of 37.5oC or or more or confirmed history of fever within previous 24 hours
* Weigh 7.5kg or over
* Screening haemoglobin (Hb) of 7g/dl or over, or haematocrit of 25% or more(If Hb not available at screening)
* Willingness to comply with the study visits and procedures, as outlined in the informed consent form
* Written or oral witnessed consent has been obtained from parent or guardian
* Assent is given by a child aged 12 years or over, in addition to the consent of their parent or guardian

Exclusion criteria:

* Features of severe/complicated falciparum malaria
* Hypersensitivity to active substances (chlorproguanil, dapsone, artesunate, artemether, lumefantrine)
* Known allergy to biguanides, sulphones, sulphonamides, artemisinin derived products or aminoalcohol drugs
* Known history of G6PD deficiency
* Infants with a history of hyperbilirubinaemia during the neonatal period
* Use of concomitant medications that may induce haemolysis or haemolytic anaemia from the WHO (World Health Organization) list of essential drugs
* Evidence of any concomitant infection at the time of presentation (including P. vivax, P. ovale and P. malariae)
* Any other underlying disease that may compromise the diagnosis and the evaluation of the response to the study medication (including clinical symptoms of immunosuppression, tuberculosis, bacterial infection; cardiac or pulmonary disease)
* Malnutrition, defined as a child whose weight-for-height is below -3 standard deviations or less than 70% of the median of the NCHS/WHO normalised reference values
* Treatment within the past three months with mefloquine or mefloquine-sulphadoxine-pyrimethamine; twenty-eight days with sulphadoxine/pyrimethamine, sulfalene/pyrimethamine, lumefantrine or artemether/lumefantrine, amodiaquine, atovaquone or atovoquone/proguanil, halofantrine; 14-days with chlorproguanil/dapsone, or 7-days with quinine (full course), proguanil, artemisinins, tetracycline doxycycline or clindamycin
* Positive sulphadoxine/pyrimethamine urine screen for 'unknown' antimalarial drug use in prior 28-days
* Use of an investigational drug within 30 days or 5 half-lives whichever is the longer
* Previous participation in this study
* Female subjects of child-bearing age, who have had a positive pregnancy test at screening, or do not give their consent to take a pregnancy test
* Female subjects who will be breast-feeding an infant for the duration of the study

Ages: 12 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1395 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Parasitological cure rate, PCR corrected, at day 28 in the PP population The ITT population is a key supportive analysis.

SECONDARY OUTCOMES:
Parasitological cure rate, PCR-corrected, at day 14 and 42 ACPR, and ACPR PCR corrected at day 14, 28 and 42 Summary of asexual parasite densities on days 0, 1, 2, 3, 7, 14, 28 and 42 by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Bobo-Dioulasso, Burkina Faso
- GSK Investigational Site, Kintampo, Ghana
- Kenya (2):
  - GSK Investigational Site, Eldoret
  - GSK Investigational Site, Kilifi
- Nigeria (4):
  - GSK Investigational Site, Barkin Ladi
  - GSK Investigational Site, Calabar
  - GSK Investigational Site, Enugu
  - GSK Investigational Site, Ibadan
- GSK Investigational Site, Ifakara, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pamba A, Richardson ND, Carter N, Duparc S, Premji Z, Tiono AB, Luzzatto L. Clinical spectrum and severity of hemolytic anemia in glucose 6-phosphate dehydrogenase-deficient children receiving dapsone. Blood. 2012 Nov 15;120(20):4123-33. doi: 10.1182/blood-2012-03-416032. Epub 2012 Sep 19. PMID 22993389
- [Derived] Carter N, Pamba A, Duparc S, Waitumbi JN. Frequency of glucose-6-phosphate dehydrogenase deficiency in malaria patients from six African countries enrolled in two randomized anti-malarial clinical trials. Malar J. 2011 Aug 17;10:241. doi: 10.1186/1475-2875-10-241. PMID 21849081
- [Derived] Premji Z, Umeh RE, Owusu-Agyei S, Esamai F, Ezedinachi EU, Oguche S, Borrmann S, Sowunmi A, Duparc S, Kirby PL, Pamba A, Kellam L, Guiguemde R, Greenwood B, Ward SA, Winstanley PA. Chlorproguanil-dapsone-artesunate versus artemether-lumefantrine: a randomized, double-blind phase III trial in African children and adolescents with uncomplicated Plasmodium falciparum malaria. PLoS One. 2009 Aug 19;4(8):e6682. doi: 10.1371/journal.pone.0006682. PMID 19690618
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CDA 714703/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register